CLINICAL TRIAL: NCT05096936
Title: Pilates Method and/or Photobiomodulation Therapy Combined to Static Magnetic Field in Women With Stress Urinary Incontinence: What is Better?
Brief Title: Pilates Method and/or Photobiomodulation in Women With Stress Urinary Incontinence
Acronym: PBMT-IUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade de Caxias do Sul (Other)
Responsible Party: Principal Investigator, Thiago De Marchi, DR, Clinical Professor, Universidade de Caxias do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBMT and IUE
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Laser Therapy; Urinary Incontinence,Stress; Pilates Method
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Exercise Movement Techniques; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates PBMT (Experimental): This group will receive training in the Pilates method associated with the effective application of photobiomodulation.
  Interventions: Other: Pilates; Other: Photobiomodulation
- Pilates (Experimental): This group will receive training in the Pilates method associated with the not effective (placebo) application of photobiomodulation.
  Interventions: Other: Pilates
- PBMT (Placebo Comparator): This group will receive effective application of photobiomodulation and will not perform the pilates method training
  Interventions: Other: Photobiomodulation

INTERVENTIONS:
Other: Pilates — The solo Pilates method will be applied twice a week for 12 weeks using the following exercises:
  20 Breaths, Double leg stretch, Single leg stretch, Leg circles, Hip lift on ball, Abdominal tightening on ball, Alternating two supports, Side bend, Side kick - side kick, Side kicks, Shell and Swan and Neck pull stretches; in the tenth session, we evolved some exercises: The saw, Swan dive, Book close series, Hip lift on the ball and Front pulls; in the eighteenth session we changed again some exercises for: Leg pull back, Rolling like a Ball, Swimming, Roll over and Leg pull front.
  Other Names: Pilates exercise; Pilates Methods
  Arms: Pilates; Pilates PBMT
Other: Photobiomodulation — Applications of FBM or placebo (MR4 ACTIVet PRO Laser Shower Portable, MRM, USA) will last for 115s and will deliver 60 J at each point. The mode of application, with the patient supine on a stretcher, with the grouping probe held stationary in contact with the skin, at a 90-degree angle, in the pubic mound and in the perineum region.
  Arms: PBMT; Pilates PBMT

SUMMARY:
The present study is a clinical intervention applied to patients with urinary incontinence, with the intention of verifying the effects of the Pilates method associated or not with photobiomodulation with static magnetic field. The sample will consist of women with stress urinary incontinence from Bento Gonçalves attended at the school clinic of Faculdade Cenecista de Bento Gonçalves.

ELIGIBILITY:
Inclusion Criteria:

* Women between 30 and 60 years old;
* Present a clinical diagnosis of SUI;
* The patient must be available at pre-scheduled times for a period of 12 weeks, with full participation;
* The participant must agree with the methodology proposed by the project and, if so, must sign the TCLE as legal proof of their participation.

Exclusion Criteria:

* Patients with urge urinary incontinence;
* Constant flow urinary incontinence and stress urinary incontinence during the gestational period (because these are possible transitory cases due to pregnancy);
* Women who have difficulty in understanding;
* Patients who have more than one absence per month during the interventions.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
decreased urinary loss | 01, 09, 17 and 24 day of intervention.
  PAD test

SECONDARY OUTCOMES:
single-digital vaginal touch | 01 and 24 day of intervention.
  Muscle strength will be assessed through the unidigital vaginal touch, applied by a "blind" evaluator, so called because she does not monitor the performance of the interventions, as well as their respective evolutions during treatment, this assessment is subjective and will be classified by the scale of Modified Oxford (scale with a score between 0-5; 0- absence of muscle response, 1- Outline of non-sustained contraction; 2- presence of small intensity contraction, but which is sustained; 3- moderate contraction, felt as an increase in intravaginal pressure, which compresses the examiner's fingers with a small cranial elevation of the vaginal wall; 4- satisfactory contraction, which squeezes the examiner's fingers with elevation of the vaginal wall towards the pubic symphysis; 5- strong contraction, firm compression of the fingers of the examiner with positive movement towards the pubic symphysis).
International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | 01 and 24 day of intervention.
  The ICIQ-SF is a questionnaire used to assess urinary incontinence, consisting of six questions that assess the frequency, severity of urinary loss and the impact of urinary incontinence on daily life, in addition to a sequence of eight self-diagnostic items, related to causes or incontinence situations that are not scored. The sum of the scores for questions three, four and five ranges from 0 to 21, and the higher the total score, the greater the severity of urinary incontinence. The impact of daily life is defined according to the score of question five; (0) not at all, (1-3) mild, (4-6) moderate, (7-9) severe, and (10) very severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Escola da Faculdade Cenecista de Bento Gonçalves Clínica Escola CNECBG, Bento Gonçalves, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knorst MR, Resende TL, Santos TG, Goldim JR. The effect of outpatient physical therapy intervention on pelvic floor muscles in women with urinary incontinence. Braz J Phys Ther. 2013 Sep-Oct;17(5):442-9. doi: 10.1590/S1413-35552012005000117. Epub 2013 Oct 21. English, Portuguese. PMID 24173346
- [Background] De Marchi T, Leal Junior EC, Bortoli C, Tomazoni SS, Lopes-Martins RA, Salvador M. Low-level laser therapy (LLLT) in human progressive-intensity running: effects on exercise performance, skeletal muscle status, and oxidative stress. Lasers Med Sci. 2012 Jan;27(1):231-6. doi: 10.1007/s10103-011-0955-5. Epub 2011 Jul 8. PMID 21739259
- [Background] Coyne KS, Zhou Z, Thompson C, Versi E. The impact on health-related quality of life of stress, urge and mixed urinary incontinence. BJU Int. 2003 Nov;92(7):731-5. doi: 10.1046/j.1464-410x.2003.04463.x. PMID 14616456
- [Background] de Almeida P, Lopes-Martins RA, De Marchi T, Tomazoni SS, Albertini R, Correa JC, Rossi RP, Machado GP, da Silva DP, Bjordal JM, Leal Junior EC. Red (660 nm) and infrared (830 nm) low-level laser therapy in skeletal muscle fatigue in humans: what is better? Lasers Med Sci. 2012 Mar;27(2):453-8. doi: 10.1007/s10103-011-0957-3. Epub 2011 Jul 22. PMID 21814736